CLINICAL TRIAL: NCT04117932
Title: Efficacy and Safety of Ustekinumab in Bullous Pemphigoid
Acronym: PB-USTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO19083
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-03

CONDITIONS: Bullous Pemphigoid
Keywords: bullous pemphigoid; ustekinumab; superpotent topical corticosteroids; efficacy; safety
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm "ustekinumab" (Experimental): Patients with bullous pemphigoid, treated using ustekinumab in association during 8 weeks with superpotent topical corticosteroids
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab (90 mg subcutaneously at weeks 0, 4, 16), in association with topical superpotent corticosteroid (10-30 g per day during the first 4 weeks, then every other day during 4 weeks).

SUMMARY:
Bullous pemphigoid (BP) is an autoimmune subepidermal blistering disease and typically affects the elderly. Clinically, BP is an intensely pruritic erythematous eruption with widespread blister formation. BP is usually a chronic disease, with spontaneous exacerbations and remissions, which may be accompanied by significant morbidity.

BP usually requires on average a 1-year duration of treatment. Superpotent topical corticosteroids have been demonstrated to be effective. Despite their high efficacy, topical corticosteroids are often considered as poorly convenient, requiring the assistance of patients' relatives or a nurse to apply the topical treatment on a long period of time.

Overall, whereas BP lesions can be adequately and rapidly controlled with either topical corticosteroids, there is a high need for a safe maintenance therapy to avoid treatment side effects due to cumulative doses of corticosteroids over months.

Newer therapeutic agents such as ustekinumab targeting molecules involved in the inflammatory cascade associated with BP represent future alternatives to classical immunosuppressant drugs for maintenance therapy.

DETAILED DESCRIPTION:
The aim of the study is to evaluate efficacy of ustekinumab in association during 8 weeks with superpotent topical corticosteroids in patients with bullous pemphigoid

ELIGIBILITY:
inclusion criteria :

* patient with bullous pemphigoid
* patient aged between 18 and 90
* patient with Karnofsky Performance score > 60%
* patient agreed to participate to the study

exclusion criteria :

* patient with allergy to corticosteroids
* patient with allergy to ustekinumab
* patient with any severe medical condition at time of inclusion including stroke, heart failure, renal failure, high blood pressure and diabetes mellitus
* malignancy < 5 years prior to inclusion
* pregnant or nursing (lactating) women, or women of child-bearing potential
* active infection or with recent history of clinically significant infection within 4 weeks prior to inclusion
* history or presence of infection with hepatitis B or C.
* history or presence of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
complete remission | 28 weeks
  Complete remission is defined as the absence of new or established lesions (bullae, eczematous lesions or urticarial lesions)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France